CLINICAL TRIAL: NCT00354913
Title: A Phase II Study of Imatinib Mesylate Plus Hydroxyurea in the Treatment of Patients With Recurrent/Progressive Meningioma
Brief Title: Imatinib Mesylate and Hydroxyurea in Treating Patients With Recurrent or Progressive Meningioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006768; DUMC-7082-05-4R0; NOVARTIS-DUMC-7082-05-4R0; NCT00611234 (obsolete NCT alias)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2013-01-14 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-12

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: adult grade I meningioma; adult grade II meningioma; adult grade III meningioma; adult papillary meningioma; adult anaplastic meningioma; recurrent adult brain tumor; glioblastoma multiforme (GBM); Imatinib; Imatinib mesylate; Hydroxyurea; Droxia; Hydrea; Hydroxycarbamide; Gleevec; Meningioma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Meningioma; Brain Neoplasms | interventions — Hydroxyurea; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib mesylate+hydroxyurea (Experimental): All patients receive imatinib mesylate and hydroxyurea orally on a daily, continuous basis. Dosing of imatinib mesylate is adjusted for patients who are also receiving p450-inducing anti-epileptic drugs.
  Interventions: Drug: hydroxyurea; Drug: imatinib mesylate

INTERVENTIONS:
Drug: hydroxyurea — Hydroxyurea is administered orally twice a day. The dose will be set at 500 mg twice a day for all patients. If vomiting occurs not additional trial medication should be taken that day in an effort to replace the material that has been vomited. It is recommended that patients take their prescribed hydroxyurea at the same time that they take their prescribed imatinib mesylate, however, a 30-60 minute interval between agents is acceptable, if required for practical or other compliance issues.
  Other Names: Droxia; Hydrea; Hydroxycarbamide
Drug: imatinib mesylate — Imatinib administered orally on daily, continuous basis. Imatinib doses of 400mg/600mg administered once daily, whereas daily doses of 800mg/greater administered as equally divided dose taken twice day.
  Dose for Imatinib:
  Patients receiving p450-inducing antiepileptic drugs:500mg twice day Patients not receiving p450-inducing antiepileptic drugs:400mg/day.
  If patients who were not on Cytochrome P450, family 3, subfamily A (CYP3A) enzyme-reducing anti-epileptic drug (EIAED) when originally enrolled must initiate CYP3A enzyme-inducing anti-epileptic drug while on study, study regimen will remain same for minimum of 2 wks before pt transitions to dosing as specified for patients on anti-epileptic drug. If patients originally enrolled must discontinue all EIAEDs while on study, in interest of patient safety, dosing of study regimen will transition to that of patients not on anti-epileptics immediately.
  Other Names: Gleevec

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as hydroxyurea, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving imatinib mesylate together with hydroxyurea may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving imatinib mesylate together with hydroxyurea works in treating patients with recurrent or progressive meningioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the activity of imatinib mesylate and hydroxyurea, as measured by 6-month progression-free survival, in patients with recurrent or progressive meningioma.

Secondary

* Evaluate the progression-free survival (PFS)
* Overall survival (OS),
* Objective response rate among patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive oral imatinib mesylate once or twice daily and oral hydroxyurea twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 21 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed meningioma
* Recurrent or progressive disease after prior surgical resection
* Measurable disease by contrast-enhanced MRI
* Multifocal disease allowed
* No evidence of intratumor hemorrhage on pretreatment diagnostic imaging

  * Stable postoperative grade 1 hemorrhage allowed
* No peripheral edema or central or systemic fluid collections ≥ grade 2 (e.g., pericardial effusion, pulmonary effusion, ascites)

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Absolute neutrophil count > 1,500/mm³
* Hemoglobin > 9 g/dL
* Platelet count > 100,000/mm³
* Potassium normal*
* Calcium normal*
* Magnesium normal*
* Phosphorus normal*
* alanine aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Creatinine < 1.5 times ULN OR creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No excessive risk of bleeding, as defined by stroke within the past 6 months
* No active systemic bleeding (i.e., gastrointestinal bleeding or gross hematuria)
* No history of central nervous system (CNS) or intraocular bleeding or septic endocarditis
* No concurrent severe and/or uncontrolled medical disease, including any of the following:

  * Uncontrolled diabetes
  * Congestive cardiac failure
  * Myocardial infarction within the past 6 months
  * Poorly controlled hypertension
  * History of labile hypertension
  * History of poor compliance with antihypertensive regimen
  * Chronic renal disease
  * Active uncontrolled infection requiring intravenous antibiotics
* No acute or chronic liver disease (i.e., hepatitis, cirrhosis)
* No HIV positivity
* No impairment of gastrointestinal function or disease that may significantly alter the absorption of imatinib mesylate, including any of the following:

  * Ulcerative disease
  * Uncontrolled nausea
  * Vomiting
  * Diarrhea
  * Malabsorption syndrome
  * Bowel obstruction
  * Inability to swallow tablets
* No other malignancy within the past 5 years except basal cell skin cancer or cervical carcinoma in situ NOTE: *Unless correctable with supplements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* More than 1 week since prior tumor biopsy
* More than 2 weeks since prior surgical resection
* Prior hydroxyurea allowed provided patient has not had progressive disease or toxicity > grade 3
* No prior imatinib mesylate or other platelet-derived growth factor-directed therapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)*

  * Chemotherapeutic agents such as etoposide that are normally given at shorter intervals allowed even if < 4 weeks from last prior dose of chemotherapy
* At least 4 weeks since prior radiotherapy*
* At least 1 week since prior biological, immunotherapeutic, or cytostatic drugs
* At least 2 weeks since prior investigational drugs
* No concurrent warfarin NOTE: *Unless there is unequivocal evidence of tumor progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-05; Primary Completion 2009-03 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

REFERENCES:
- [Result] Reardon DA, Norden AD, Desjardins A, Vredenburgh JJ, Herndon JE 2nd, Coan A, Sampson JH, Gururangan S, Peters KB, McLendon RE, Norfleet JA, Lipp ES, Drappatz J, Wen PY, Friedman HS. Phase II study of Gleevec(R) plus hydroxyurea (HU) in adults with progressive or recurrent meningioma. J Neurooncol. 2012 Jan;106(2):409-15. doi: 10.1007/s11060-011-0687-1. Epub 2011 Sep 22. PMID 21938530

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imatinib Mesylate+Hydroxyurea
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate+Hydroxyurea
Number analyzed (Participants) | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 54.0 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months
Description: Percentage of participants surviving six months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression according to the Macdonald criteria, or death due to any cause.
Time Frame: From the date of study treatment initiation to the date of the first documented progression or death from any cause, whichever came first, assessed up to 69 months. For each participant, PFS was assessed at 6 months after treatment initiation.
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imatinib Mesylate+Hydroxyurea
Number analyzed (Participants) | 21
percentage of participants | 61.9 [38.1 to 78.8]

2. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression according to Macdonald criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Time Frame: From the date of study treatment initiation to the date of the first documented progression or death from any cause, whichever came first, assessed up to 69 months.
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib Mesylate+Hydroxyurea
Number analyzed (Participants) | 21
months | 7 [3.8 to 9.2]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Time in months from the start of study treatment to date of death due to any cause. Patients alive at last follow-up are censored as of that follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: From the date of study treatment initiation to the date of death from any cause, assessed up to 69 months.
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib Mesylate+Hydroxyurea
Number analyzed (Participants) | 21
months | 66 [20.7 to 66]

4. Secondary Outcome: Objective Response Rate
Description: Percentage of participants with an objective response (complete response or partial response). Per modified Macdonald criteria and assessed by MRI, complete response (CR) was the disappearance of all target lesions and partial response (PR) was a ≥50% decrease in the sum of the longest diameter of target lesions. Objective response = CR+PR.
Time Frame: 69 Months
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Imatinib Mesylate+Hydroxyurea
Number analyzed (Participants) | 21
percentage of participants | 0

ADVERSE EVENTS:
Description: Adverse Events were gathered in Common Terminology Criteria for Adverse Events (CTCAE) v. 3.0 and converted to CTCAE v. 4.0 for entry into ClinicalTrials.gov
Arm/Group | Imatinib Mesylate+Hydroxyurea
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate+Hydroxyurea (N=21)
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate+Hydroxyurea (N=21)
Anemia (Blood and lymphatic system disorders) | 5
Blurred Vision (Eye disorders) | 4
Extraocular muscle paresis (Eye disorders) | 1
Eye disorders-Other, Inflammation: right eye (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Vitreous hemorrhage (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Gastrointestinal disorders-Other: increased Appetite (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Rectal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 4
Non-cardiac chest pain (General disorders) | 1
Infections and infestations-Other: ear drainage (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Investigations-Other: BUN, high (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 3
Weight gain (Investigations) | 1
White blood count decreased (Investigations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Ataxia (Nervous system disorders) | 2
Cognitive disturbance (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysphasia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Memory impairment (Nervous system disorders) | 3
Nervous systems disorders-Other: gait (Nervous system disorders) | 1
Nervous system disorders-Other: Mood Alteration NOS (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Psychosis (Psychiatric disorders) | 1
Renal and urinary disorders-Other: nocturia (Renal and urinary disorders) | 1
Reproductive system and breast disorders-Other: NOS (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes